CLINICAL TRIAL: NCT02261324
Title: Is the Four Metre Gait Speed a Useful Outcome Measure in Patients With Acute Myocardial Infarction After Primary Percutaneous Coronary Intervention?
Brief Title: Is the 4MGS a Useful Outcome Measure Post-PPCI
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2013LF001H
Record Dates: First submitted 2014-05-01; First posted 2014-10-10 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Acute Myocardial Infarction
Keywords: Percutaneous coronary intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study aims to assess usual walking speed (4-metre gait speed) in patients undergoing primary percutaneous coronary intervention (PCI) for acute myocardial infarction and to assess whether this can predict future cardiovascular events and death.

ELIGIBILITY:
Inclusion Criteria:

* Any patient hospitalised with an acute myocardial infarction who has undergone primary percutaneous coronary intervention
* Capacity to consent
* Able to walk
* Age over 18 years

Exclusion Criteria:

* Significant co-morbidities that would limit exercise capacity or make exercise unsafe (e.g. neuromuscular disease, severe hip/lower limb joint pain, peripheral vascular disease, lower limb amputation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient hospitalised for primary percutaneous coronary intervention for acute myocardial infarction. The cohort will be recruited from Harefield hospital
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2013-12; Primary Completion 2017-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 1 year

SECONDARY OUTCOMES:
Occurrence of cardiovascular events | 1 and 5 years
Need for repeat revascularisation | 1 and 5 years
Health resource usage | 1 and 5 years
All-cause mortality | 5 years
Cardiovascular death | 1 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: William DC Man, FRCP PhD, Principal Investigator — NIHR Respiratory Biomedical Research Unit Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Harefield Hospital, Harefield, Middlesex, United Kingdom